CLINICAL TRIAL: NCT02824406
Title: Cerebrovascular Reserve Measurements in Sickle Cell Disease: an MRI Study
Brief Title: Cerebrovascular Reserve Measurements in Sickle Cell Disease
Acronym: CRUISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, B.J. Biemond, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: CRUISE study
Record Dates: First submitted 2016-02-09; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Anemia; Cerebrovascular Reserve; Perfusion; Vasculopathy; Magnetic Resonance Imaging
MeSH Terms: conditions — Anemia, Sickle Cell; Vascular Diseases | interventions — Acetazolamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The following outcomes will be assessed from veinous-drawn blood samples: Sodium, Potassium, Creatinine, Bilirubin, ASAT(SGOT), ALAT (SGPT), LDH, Ferritin, Haptoglobin, Hemoglobin, Erythrocytes, Leukocytes, Thrombocytes, MCV, MCH, MCHC, RDW, Hemoglobin, Hematocrit, Hb-F, Hb-A2, Hb-S, Hb-A2, Reticulocytes, Lymphocytes, ADAMTS13, D-Dimer, von Willebrand activity / antigen / multimer, hs-CRP, F1+2, PAI-1 antigen, t-PA-Ag antigen, NETs, Circulating histones, Metalloproteinase, Interleukin 6,13 and 18, Free HB, ADMA asymmetric dimethylarginine, VCAM, ICAM, AGEs:Pentosidine, CML - carboxyl methyl lysine, Thrombospondin, GFAP, L-selectin, VEGF, Pentraxine-3
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: CVR assessment consists of CBF measurement with arterial spin labelling (ASL)-MRI before and after intravenous administration of 16mg/kg acetazolamide (Diamox)
  Interventions: Drug: Acetazolamide
- Controls: CVR assessment consists of CBF measurement with arterial spin labelling (ASL)-MRI before and after intravenous administration of 16mg/kg acetazolamide (Diamox)
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide is administered to all participants to induce vasodilation, in order to assess the physiologic response on cerebral blood flow.
  Other Names: Diamox

SUMMARY:
The primary aim of this study is to evaluate MRI-based cerebrovascular reserve (CVR) measurements in adult patients with Sickle Cell Disease (SCD).

The primary objective is to assess whether there is a correlation between CVR and silent cerebral infarcts (SCIs).

DETAILED DESCRIPTION:
CVR is hypothesized to be impaired in SCD patients and could account for the white matter hyperintensities seen on MRI in these patients. Cerebral blood flow (CBF) alone is not sufficient to provide insight into the hemodynamic status of the brain. CVR allows us to gain insight into the capacity of the cerebrovasculature to respond to increased CBF. Vasculopathy is common in SCD and the caliber of the vessels can be assessed with 4D Flow MRI in response to actue and chronic changes in the velocity and wall shear stress on the intracranial arteries in the Circle of Willis.

This study will be performed as a single center, patient-control, cross-sectional, observational study in patients with steady-state SCD and controls. The investigators expect that patients with impaired CVR will have a greater number and/or volume of SCIs.

ELIGIBILITY:
Inclusion Criteria Patient group:

* Sickle cell disease; either homozygous sickle cell disease (HbSS), or HbSβ0 thalassemia
* 18 years of age or older
* Informed consent

Inclusion Criteria Control group:

* Similar ethnic background as Patient group
* 18 years of age or older
* Informed consent

Exclusion Criteria Patient group and Control group:

* Inability of the patient to provide informed consent or legally incompetent/incapacitated to do so
* Contraindications for MRI, such as pregnancy, claustrophobia or the presence of metal in the body
* Sickle cell crisis at the moment of participation
* History of cerebral pathology that compromises measurements, such as cerebral palsy, brain tumour,meningitis, overt infarct
* Brain surgery performed in the last 3 months
* Severe liver, heart or renal dysfunction (clearance < 10 mL/min)
* Allergy to sulphonamide
* Breastfeeding
* Use of phenytoin, procaine or acetylsacylic acid ("Ascal/aspirin")
* Risk of hypokalaemia (use of diuretics, primary hyperaldosteronism)
* Addison's Disease
* Severe asthma or emphysema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are eligible if they have a diagnosis of sickle cell disease; either homozygous sickle cell disease (HbSS), or HbSβ0 thalassemia and are in a steady disease state i.e. no crisis requiring hospitalization 4 weeks prior to participation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular Reserve (CVR) from arterial spin labelling-MRI in patients compared to controls | 20 minutes
  Cerebral blood flow (CBF mL/100g/min) measurement before, during, and after, an intravenous administration of 16mg/kg acetazolamide. The percentage change in CBF will be used as a measure for CVR (%).

SECONDARY OUTCOMES:
Cerebral Metabolic Rate of Oxygen in patients and controls | 2 minutes
  Oxygen extraction fraction and cerebral blood flow are proportional to the cerebral metabolic rate of oxygen. Using the CBF from the primary outcome, and having measured the T2 of blood (which is dependent on oxygen), we can derive the oxygen extraction fraction, which allows us to calculate the cerebral metabolic rate of oxygen (CMRO2) and compare patients with controls.
Blood markers relating to anemia will be related to MRI findings | Through study completion, an average of 1 year
  Hematocrit, hemoglobin, hemolysis, red blood cell count, mean corpuscular hemoglobin concentration.
Velocity in the circle of willis assessed with 4D Flow MRI | 10 minutes
  Velocity (m/s) before and after acetazolamide challenge will be used to indicate cerebrovascular reserve and compared between patients and controls
Silent Cerebral Infarct (SCI) on T2-weighted FLAIR MRI | 10 minutes
  Volume of SCIs will be assessed in relation to CVR

CONTACTS AND LOCATIONS:
Overall Officials: AJ Nederveen, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes